CLINICAL TRIAL: NCT05672134
Title: Evaluation of GeranylGeranylAcetone in Heart Failure With Preserved Ejection Fraction
Acronym: GLADIATOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M. Louis Handoko, MD, PhD, Principal investigator, VU University of Amsterdam
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL 80684
Record Dates: First submitted 2022-06-08; First posted 2023-01-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — geranylgeranylacetone; Echocardiography; Electrocardiography

STUDY DESIGN:
Intervention Model Description: crossover multi-centre, double-blind, randomized control trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Patients will receive 13 weeks of experimental treatment, followed by a 7 week wash-out period, continuing with 13 weeks of placebo as per crossover design.
  Interventions: Diagnostic Test: Iohexol measurement; Drug: Geranylgeranylacetone (GGA); Diagnostic Test: Echocardiography; Diagnostic Test: 6-minute walking distance test; Diagnostic Test: EndoPAT; Diagnostic Test: Para-amino Hippuric Acid test; Diagnostic Test: Electrocardiogram
- Placebo arm (Placebo Comparator): Patients will receive 13 weeks of placebo treatment, followed by a 7 week wash-out period, continuing with 13 weeks of experimental treatment as per crossover design.
  Interventions: Diagnostic Test: Iohexol measurement; Drug: Geranylgeranylacetone (GGA); Diagnostic Test: Echocardiography; Diagnostic Test: 6-minute walking distance test; Diagnostic Test: EndoPAT; Diagnostic Test: Para-amino Hippuric Acid test; Diagnostic Test: Electrocardiogram

INTERVENTIONS:
Diagnostic Test: Iohexol measurement — Invasive renal hemodynamic measurement of mGFR through the administration of Iohexol.
Drug: Geranylgeranylacetone (GGA) — 13 weeks of treatment with GGA/placebo orally, followed by a wash-out period of 6 weeks, then reversal of the treatment arms.
Diagnostic Test: Echocardiography — The investigators will perform echocardiography to find changes in cardiac function.
Diagnostic Test: 6-minute walking distance test — 6 minute walking distance test to compare exercise tolerance in participants.
Diagnostic Test: EndoPAT — Use of EndoPAT to measure endothelial function.
Diagnostic Test: Para-amino Hippuric Acid test — PAH-measurement to measure ERPF.
Diagnostic Test: Electrocardiogram — 12-lead Electrocardiogram

SUMMARY:
The goal of this double-blind randomized, placebo-controlled cross-over trial is to evaluate the effectiveness of GerenylGeranylAcetone (GGA) in patients with Heart Failure with a preserved ejection fraction.

The main questions it aims to answer are:

* What is the effect of GGA on diastolic function?
* What is the effect of GGA on endothelial function?

Main study tasks:

* Participants will be treated with either GGA or placebo for 13 weeks. After this they will have a break (wash-out) period for 6 weeks and then cross over to the other study arm.
* Cardiac function will be measured using echocardiogram in all participants
* Renal measurements and endothelial measurements will be performed on the participants.
* Participants will perform a 5 minute walking distance test for functional capacity.
* Participants will fill out questionnaires to score signs & symptoms.

Researchers will compare the patients to themselves to see if the drug improves diastolic- and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 50 years
2. Patients with a diagnosis of symptomatic chronic heart failure (New York Heart Association class II or III) AND preserved systolic LV function (LV ejection fraction or LVEF ≥ 50%) documented within the last 6 months AND evidence of diastolic LV dysfunction with at least 1 out of the following 4 criteria:

   * HFA-PEFF score ≥5
   * H2FPEF score ≥6
   * HFpEF according to the 2021 ESC HF Guidelines (NT-proBNP>125 pg/ml AND either LV mass indexed or LVMI >95 g/m2 for women and >115 g/m2 for men OR left atrial volume indexed or LAVI >34 ml/m2 OR mean e; septal/lateral < 9 cm/s) OR E/e' >13 OR TR velocity at rest >2,8m/s.
   * Pulmonary capillary wedge pressure (PCWP) >15 mmHg and/or >25 mmHg during exercise.

Exclusion Criteria:

1. Current acute decompensated heart failure, requiring hospitalization or augmented therapy with intravenous diuretics, vasodilators, and/or inotropic drugs
2. Acute coronary syndrome, transient ischemic attack/cerebrovascular accident, major surgery within the previous 3 months
3. Hemoglobin <9 g/dl at screening
4. LVEF <40% measured at any time point in the history of the patient
5. History of mitral valve repair or replacement
6. Presence of significant valvular disease defined as mitral valve regurgitation defined as grade ≥ 3+ MR; tricuspid valve regurgitation defined as grade ≥ 2+ TR; aortic valve disease defined as ≥ 2+ AR or > moderate AS
7. Acute myocarditis within 3 months prior to randomization
8. Infiltrative cardiomyopathy
9. Genetic cardiomyopathy
10. Severe pulmonary disease requiring home oxygen or chronic oral steroid therapy
11. Precapillary pulmonary hypertension
12. BMI >40 kg/m2
13. Estimated glomerular filtration rate (GFR) <20 ml/min or >90 ml/min
14. History of solid organ transplantation including kidney transplantation
15. Atrial fibrillation or atrial flutter with resting ventricular rate >110 bpm
16. Not able to undergo the complete study protocol
17. Doubt about compliance
18. Pre-menopausal women who are nursing, pregnant, or of child-bearing potential and not practicing an acceptable method of birth control
19. Chronic absorption problems
20. Proven allergy for lactose products or cow-milk.
21. Proven allergy for Iodide-containing contrast, Iohexol or PAH.
22. Any documented or suspected malignancy or history of malignancy within 1 year prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix
23. Currently enrolled in another investigational device or drug trial
24. Estimated life expectancy <1 year

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Filling pressures | after 13 weeks of treatment
  Changes in echocardiography determined filling pressures (E/e')?
Endothelial function | after 13 weeks of treatment
  Changes in EndoPAT®-derived reactive hyperemia index (RHI)

SECONDARY OUTCOMES:
Left atrial volumes | After 13 weeks of treatment
  Changes in echogardiographic measured left atrial volume index (LAVI)
Left atrial global strain | After 13 weeks of treatment
  Changes in echogardiographic measured LA global strain (LAGS)
Left atrial emptying fractions | After 13 weeks of treatment.
  Changes in echogardiographic LA emptying fractions. Formula: (LA maximum volume-LA minimum volume)/LA maximum volume × 100%
Left Ventricular global longitudinal strain | Ater 13 weeks of treatment
  Changes in echocardiographically determinded LV global longitudinal strain (LGS)
Left Ventricular Myocardial relaxation | Ater 13 weeks of treatment
  Change in echocardiographically determined myocardial relaxation (e')
Left Ventricular distensibility | After 13 weeks of treatment
  Change in echocardiographically determined LV distensibility, measured by E.
Right Ventricular systolic function | After 13 weeks of treatment
  Change in echocardiographically determined RV TAPSE
Pulmonary Artery Pressure | After 13 weeks of treatment
  Change in echocardiographically determined PAP
Patient reported symptoms | After 13 weeks of treatment
  Evaluation of symptoms using New York Heart Association class (NYHA)
Quality of life assessment | After 13 weeks of treatment.
  Evaluation of quality of life using the Kansas City Cariomyopathy Questionnaire
Functional capacity | After 13 weeks of treatment.
  Evaluation of Functional Capacity using 6-minute walking distance test (6MWD)
CRP (inflammatory biomarker) | After 13 weeks of treatment
  Changes in CRP concentration in serum
Nitrosated hemoglobin (microvascular marker) | After 13 weeks of treatment
  Changes in Nitrosated hemoglobin (Hb(NO)4) concentration in serum
Nitrate (microvascular marker) | After 13 weeks of treatment
  Changes in nitrate concentration in serum
Endothelin-1 (microvascular marker) | After 13 weeks of treatment
  Changes in Endothelin-1 concentration in serum
H2S (microvascular marker) | After 13 weeks of treatment
  Changes in H2S concentration in serum
Measured Glomerular Filtration Rate (mGFR) | After 13 weeks of treatment
  Changes in mGFR using Iohexol measurements in urine
Effective Renal Plasma Flow (ERPF) | After 13 weeks of treatment
  Changes in ERPF using PAH-measurements in urine
Renal vascular resistance (RVR) | After 13 weeks of treatment
  Changes in intrakidney hemodynamic function (Systemic Blood pressure / Renal Blood Flow)
Urine Albumine Creatinin Ratio | After 13 weeks of treatment
  Changes in UACR concentration measured in urine.
Neutrophil gelatinase associated lipocalin (NGAL) | After 13 weeks of treatment
  Changes in NGAL concentration measured in urine and serum
Kidney Injury marker 1 (KIM-1) | After 13 weeks of treatment
  Changes in KIM-1 concentration measured in urine and serum

OTHER OUTCOMES:
N-terminal pro Brain Natriuretic Peptide (NT-proBNP) | After 13 weeks of treatment
  Changes in NT-proBNP measured in serum
Troponin T | After 13 weeks of treatment
  Changes in Troponin T measured in serum
Clinical events | After 13 weeks of treatment
  Comparison of the frequency of a combined safety endpoint of death, myocardial infarction and heart failure hospitalization
Serious Adverse Events (SAE's) | After 13 weeks of treatment.
  Comparison of the frequency of Serious Adverse Events between both groups.
Treatment Emergent Adverse Events (TEAE's) | After 13 weeks of treatment.
  Comparison of the frequency of Treatment Emergent Adverse Events between both groups.
Adverse events of specific interest (AESI's) | After 13 weeks of treatment
  Comparison of the frequency of Adverse events of specific interest between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Handoko, MD, PhD, Principal Investigator — Amsterdam University Medical Center; Adriaan Voors, MD, PhD, Principal Investigator — University Medical Center Groningen; Loek van Heerebeek, MD, PhD, Principal Investigator — Onze Lieve Vrouwe Gasthuis, Amsterdam
Locations (1):
- Amsterdam UMC, loc VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No